CLINICAL TRIAL: NCT05401760
Title: Combined Phacoaspiration and Angle Surgery Versus Phacoaspiration in Pediatric Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina abdelfattah, lecturer of ophthalmology Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.22.05.1718
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  1. Patients with pediatric congenital cataract Aged less than two years associated with other ocular anomalies which is high risk for developing PCSG as microcornea and aniridia.
  2. Patient with pediatric cataract with other eye had post cataract surgery glaucoma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: includes eyes for whom combined phacoaspiration & angle surgery will be done. (Active Comparator): Group A: for whom combined phacoaspiration & angle surgery trabeculotomy will be done.
  * continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
  * The nucleus and cortex will be aspirated.
  * Posterior capsulrehxis and limited anterior vitrectomy will be done.
  * Corneal incisions will be sutured with 10-0 Nylon suture.
  * Using metal trabeculotomes to open thetrabecular meshwork after accessing the canal of schlemm.
  * Suturing of scleral flap with 10-0 Nylon suture.
  Interventions: Procedure: Group A :combined phacoaspiration and angle surgery
- Group B : includes eyes with only phacoaspiration will be done (Active Comparator): Group B: for whom phacoaspiration only will be done.
  * 2 side ports will be fashioned.
  * Trypan blue will be injected to aid visualization of the anterior capsule & continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
  * The nucleus and cortex will be aspirated.
  * Posterior capsulrehxis and limited anterior vitrectomy will be done.
  * Corneal incisions will be sutured with 10-0 Nylon suture.
  Interventions: Procedure: Group B : phacoaspiration only

INTERVENTIONS:
Procedure: Group A :combined phacoaspiration and angle surgery — * Partial thickness scleral flap to access the canal of schlemm.
  * 2 side ports will be fashioned.
  * Trypan blue will be injected to aid visualization of the anterior capsule & continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
  * The nucleus and cortex will be aspirated.
  * Posterior capsulrehxis and limited anterior vitrectomy will be done.
  * Corneal incisions will be sutured with 10-0 Nylon suture.
  * Using metal trabeculotomes to open thetrabecular meshwork after accessing the canal of schlemm.
  * Suturing of scleral flap with 10-0 Nylon suture.
  Arms: Group A: includes eyes for whom combined phacoaspiration & angle surgery will be done.
Procedure: Group B : phacoaspiration only — * 2 side ports will be fashioned.
  * Trypan blue will be injected to aid visualization of the anterior capsule & continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
  * The nucleus and cortex will be aspirated.
  * Posterior capsulrehxis and limited anterior vitrectomy will be done.
  * Corneal incisions will be sutured with 10-0 Nylon suture.
  Arms: Group B : includes eyes with only phacoaspiration will be done

SUMMARY:
The aim of this study is to report the effectiveness of phacoaspiration when combined with angle surgery in preventing postoperative glaucoma following pediatric cataract surgery

DETAILED DESCRIPTION:
As postoperative glaucoma could be the consequence of a dysgenesis of the iridocorneal angle that accompanies the dysgenesis of the lens so, the hypothesis states that combined phacoaspiration with angle surgery may be superior to phacoaspiration as standalone procedure in controlling IOP within the normal range postoperatively after pediatric cataract surgery

• Patients with pediatric cataract will be subdivided into 2 groups: Group A: includes eyes for whom combined phacoaspiration & angle surgery will be done.

Group B: includes eyes for whom phacoaspiration only will be done. All surgeries will be performed in Mansoura Ophthalmic Center by the same surgeon or under his supervision.

Preoperative:

1. History: Full ocular & general history will be taken Ocular history: history of ocular trauma, ocular surgeries & wearing glasses. General medical history: age, history of any associated neurologic, metabolic or systemic disease or drug intake.
2. Examination: Full ocular examination will be done

   * Anterior segment examination using (Topcon or Zeiss surgical microscopes) or (Zeiss or hag streit slit lamps).
   * Corneal diameter will be measured.
   * Fundus examination using indirect ophthalmoscope (KEELER Vantage Plus indirect ophthalmoscope) if the fundus is visible.
   * IOP measuring using Schoitz tonometer.
   * Refraction (if the eye can be refracted) & K readings will be measured using portable autorefractometer (Retinomax K-plus2).
3. Investigations:

   * Axial length, anterior chamber depth & Ocular biometry will be measured using (Nidek Al-Scan Optical Biometer).
   * B-scan will be done using (Nidek Us-4000 Echoscan).
   * Ultrasound biomicroscopy (UBM) scan will be performed using (VuMAX HD).

Intraoperative:

1. Group A: for whom combined phacoaspiration & angle surgery ither trabeculotomy will be done. I

   * Partial thickness scleral flap to access the canal of schlemm.
   * 2 side ports will be fashioned.
   * Trypan blue will be injected to aid visualization of the anterior capsule & continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
   * The nucleus and cortex will be aspirated.
   * Posterior capsulrehxis and limited anterior vitrectomy will be done.
   * Corneal incisions will be sutured with 10-0 Nylon suture.
   * Using metal trabeculotomes to open thetrabecular meshwork after accessing the canal of schlemm.
   * Suturing of scleral flap with 10-0 Nylon suture.
2. Group B: for whom phacoaspiration only will be done.

   * 2 side ports will be fashioned.
   * Trypan blue will be injected to aid visualization of the anterior capsule & continuous curvilinear anterior capsulorhexis of approximately 5.0 mm diameter will be done.
   * The nucleus and cortex will be aspirated.
   * Posterior capsulrehxis and limited anterior vitrectomy will be done.
   * Corneal incisions will be sutured with 10-0 Nylon suture.

Postoperative:

1. All patients will be discharged on:

   * Systemic &topical antibiotic eye drops.
   * Topical steroids.
   * Cycloplegic eye drops.
   * Combined antibiotic and steroid eye ointment.
2. Topical Steroids & cycloplegic eye drops will be gradually withdrawn over a period of 3 months.
3. The eyes will be carefully examined at each follow-up visit (1 week, 2 weeks 1months and 3 months).
4. During each visit:

   * Anterior segment examination will be done.
   * Measuring of:

     * Corneal diameter.
     * Cup/disc ratio.
     * IOP using Schoitz tonometer.
     * Axial length, anterior chamber depth.

ELIGIBILITY:
Inclusion criteria:

* pediatric congenital cataract Aged less than two years associated with other ocular anomalies which is high risk for developing glaucoma as microcornea and aniridia.
* pediatric cataract with other eye had post cataract surgery glaucoma

Exclusion criteria:

* Acquired cataracts secondary to trauma or uveitis.
* Aged more than two years.
* Associated corneal opacities.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | up to one year follow up
  glaucoma

SECONDARY OUTCOMES:
rate of complications | one year follow up
  hyphaema or intraocular inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Dina Abd Elfattah, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
results of collected data